CLINICAL TRIAL: NCT02435472
Title: A Randomized Clinical Trial of Exercise vs. Usual Care Among Men Opting for Active Surveillance for Prostate Cancer
Brief Title: Active Surveillance Exercise Clinical Trial
Acronym: ASX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 135512; 1R01CA181802 (NIH); NCI-2015-01133 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-04-16; First posted 2015-05-06 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Localized Prostate Cancer; Active Surveillance for Prostate Cancer
Keywords: Active Surveillance; Exercise; Prostate cancer; Life style; Survey; Personalized exercise; Exercise trainer
MeSH Terms: conditions — Motor Activity; Prostatic Neoplasms | interventions — Exercise; Exercise Test; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: Exercise (Experimental): Arm A will engage in up to 4 aerobic sessions per week at 55% to 75% of the individually determined exercise capacity (VO2peak; determined from the cardiopulmonary exercise test (CPET) performed at baseline) for 16 weeks. This exercise prescription will be achieved through ~ 4 sessions / week. Men are provided with a heart rate monitor to help ensure they exercise in their target zone. At baseline & week 16, all patients will complete: (1) lifestyle and quality-of-life questionnaires, (2) measurement of weight (3) collection of research fasting blood sample, (4) collection of urine sample, and (5) cardiorespiratory fitness testing. Archival biopsy tissue samples from before and after the intervention will also be requested.
  Interventions: Behavioral: Exercise; Other: Cardiopulmonary Exercise Test (CPET)
- Arm B: Usual Care (No Intervention): Arm B will receive print material with physical activity guidance which includes general physical activity information (e.g., "Moving through Cancer - A Guide to Exercise for Cancer Survivors") at baseline, but no specific exercise program or goals. At the conclusion of the 16 weeks, subjects in this group will be provided with a heart rate monitor, an individualized aerobic exercise program based on their cardiorespiratory fitness test results, and opportunity to consult with study exercise physiologist (one-time).
- Arm C: Exploratory (Active Comparator): Arm C is a non-randomized control group of men without cancer, which will receive all baseline and 16 week follow-up assessments (except tissue procurement) will engage in up to 4 aerobic sessions per week at 55% to 75% of the individually determined exercise capacity (VO2peak; determined from the cardiopulmonary exercise test performed at baseline) for 16 weeks. This exercise prescription will be achieved through ~ 4 sessions / week. Men are provided with a heart rate monitor to help ensure they exercise in their target zone. At baseline & week 16, all patients will complete: (1) lifestyle and quality-of-life questionnaires, (2) measurement of weight (3) collection of research fasting blood sample, (4) collection of urine sample, and (5) cardiorespiratory fitness testing.
  Interventions: Behavioral: Exercise; Other: Cardiopulmonary Exercise Test (CPET)
- Observational Non-Randomized Group (Active Comparator): There is also a non-randomized observational component to the study where biospecimens and survey data will be collected and one CPET will be administered. Individuals who will be enrolled to this group include those who do not meet all eligibility criteria for the RCT, or those who do not wish to be in a RCT, but are interested to participate in some lifestyle research.
  Interventions: Other: Cardiopulmonary Exercise Test (CPET)

INTERVENTIONS:
Behavioral: Exercise — This open-label, two-arm randomized controlled trial (RCT) will investigate the effects of 16 weeks of structured aerobic training, relative to usual care (print material with physical activity guidance) in 76 men with histologically confirmed low-risk prostate adenocarcinoma on active surveillance. The only investigational therapeutic agent being tested in this trial is a behavioral intervention in the form of aerobic training.
  Arms: Arm A: Exercise; Arm C: Exploratory
Other: Cardiopulmonary Exercise Test (CPET) — Exercise capacity test to assess peak oxygen consumption (VO2peak)
  Other Names: CPET
  Arms: Arm A: Exercise; Arm C: Exploratory; Observational Non-Randomized Group

SUMMARY:
This phase 2, open-label, dual-center, two-arm randomized controlled trial (RCT) investigates the effects of 16 weeks of structured aerobic training, relative to usual care (print material with physical activity guidance). Prostate genomic signatures represent the functional activity of all genes in the genome and are converted into genomic risk scores which correspond to the probability of a progression event (chance of having more aggressive disease). A structured exercise program may alter the genomic risk score and improve prediction of aggressive disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of remotely monitored, tailored aerobic training, compared to usual care (print material with physical activity guidance), on cardiopulmonary fitness in men on active surveillance for low-risk prostate cancer.

SECONDARY OBJECTIVES:

I. To determine the effect of aerobic training, compared with usual care, on prostate genomic signatures that predict risk of prostate cancer progression or aggressive disease; and messenger ribonucleic acid (mRNA) expression patterns in tumor and surrounding stromal (normal) tissue.

II. To determine the effect of aerobic training, compared with usual care, on patient-reported outcomes including active surveillance-specific anxiety, stress, & adherence.

III. To procure blood, urine and paraffin embedded prostate tissue for future exploratory studies.

IV. To conduct correlative science examining associations between measures of cardiopulmonary fitness, clinical features, and biomarkers of prognosis.

V. To evaluate and compare circulating and urinary biomarkers (e.g., metabolomics, proteomics) among men in Arms A, B, and C.

OUTLINE: This study is a randomized controlled trial of 16-weeks aerobic exercise (home-based walking) versus (vs.) usual care among 64 men with prostate cancer on active surveillance. There is also a non-randomized observational component to the study where we will collect biospecimens, survey, data, and administer one cardiopulmonary exercise test (CPET).

ARM A: Patients undergo structured aerobic training comprising four treadmill walking sessions a week at 55% to 75% of the individually determined exercise capacity for 16 weeks. Men are provided with a heart rate monitor to help ensure they exercise in their target zone. At baseline & week 16 (-7, +7 days), all patients complete: (1) lifestyle and quality-of-life questionnaires, (2) measurement of weight and waist circumference (3) collection of research fasting blood sample, (4) transrectal ultrasound-guided clinical biopsy, and (5) cardiorespiratory fitness testing. Archival tissue specimens from standard of care biopsies are also collected, pre/post intervention.

ARM B (USUAL CARE): Patients undergo usual care and are provided with general physical activity information ("Moving through Cancer-A Guide to Exercise for Cancer Survivors") at baseline. At the conclusion of the 16 weeks, subjects in this group will be provided with a free session with an exercise physiologist and an individualized aerobic exercise program based on their cardiorespiratory fitness test results. Archival tissue specimens from standard of care biopsies are also collected, pre/post intervention.

ARM C (NON-RANDOMIZED CONTROL GROUP): Control group of men without cancer, with a lower baseline fitness level (assessed as part of screening), who will receive all baseline and 16 week follow-up assessments (except tissue procurement), and the same intervention as Arm A. Subjects undergo structured aerobic training comprising four treadmill walking sessions a week at 55% to 75% of the individually determined exercise capacity for 16 weeks. Men are provided with a heart rate monitor to help ensure they exercise in their target zone. At baseline & week 16 (-7, +7 days), all patients complete: (1) lifestyle and quality-of-life questionnaires, (2) measurement of weight and waist circumference (3) collection of research fasting blood sample, (4) cardiorespiratory fitness testing.

OBSERVATIONAL GROUP (NON-RANDOMIZED): Biospecimens, survey, data, and administer one CPET will be collected. Individuals who will be enrolled to this group include those who do not meet all eligibility criteria for the RCT, or those who do not wish to be in a RCT, but are interested to participate in some lifestyle research.

After completion of study, patients in Arms A & B are followed up at 16 weeks, 12 months, and 24 months. Non-randomized participants (Arm C) are followed-up at 16 weeks, and Observational study participants are asked to complete surveys at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria

ARM A and ARM B:

* Histologically-documented localized (stage < T3) prostate adenocarcinoma
* Patient has selected active surveillance as their management strategy for low- or low-intermediate risk prostate cancer as defined below
* >= 10 core prostate biopsy completed prior to randomization with Gleason sum =< 6 with no pattern 4, or Gleason 3+4 in < 34% of all cores
* Diagnostic or most recent prostate specific antigen (PSA) =< 15 ng/ml, or PSA density (PSAD) < 0.15
* Low to moderate fitness level at baseline (to be assessed via interview with the exercise staff and through the CPET)
* Clearance based on medical chart review and normal electrocardiogram (ECG) (administered by a trained health professional) to undergo a symptom-limited cardiopulmonary exercise test and aerobic training intervention
* Able to achieve and complete an acceptable cardiopulmonary exercise test defined as follows: achieving peak or plateau in oxygen consumption concurrent with increased power output; a respiratory exchange ratio >= 1.1 or volitional exhaustion-rating of perceived exertion > 19
* English-speaking
* A priori, we will allow men with concurrent benign prostatic hyperplasia (prostate volume > 50 g) to have a PSA between 10-15 ng/ml; and include men with low volume Gleason 3+4 disease, because such men have similar outcomes on active surveillance to those with Gleason =< 3+3; also a priori, we will allow men with < than a 10 core biopsy at the discretion of the urologist if s/he classifies the patient as "low-risk" and a good candidate for active surveillance based on other favorable features (e.g., tumor molecular tests, prostate imaging, etc.)

NON-CANCER CONTROL GROUP (EXPLORATORY ARM C):

* Healthy males age 20-35 or >=60 yrs.
* No history of prostate cancer or other cancer.
* Medical clearance based on medical chart review and normal ECG (administered by a trained health professional) to undergo a symptom-limited cardiopulmonary exercise test and aerobic training intervention OR medical clearance based on medical chart review and sub-maximal exercise testing for the remote aerobic training intervention.
* English-speaking.
* Low to moderate fitness level at baseline (to be assessed via interview with the exercise staff and through the CPET; similar to Arms A and B); subjects will be frequency-matched to subjects in the prostate cancer exercise intervention group (Arm A) to have a similar distribution of body mass index and facilitate comparisons between these two groups.

NON-RANDOMIZED OBSERVATIONAL COMPONENT ELIGIBILITY:

* Histologically-documented localized (stage < T3) prostate adenocarcinoma.
* Undergoing or initiating active surveillance.
* Medical clearance based on medical chart review and normal ECG (administered by a trained health professional) to undergo a symptom-limited cardiopulmonary exercise test and aerobic training intervention.
* English-speaking.

Exclusion Criteria

* Any prior or concurrent treatment for prostate cancer
* Use of finasteride or dutasteride within 3 weeks or 6 months, respectively, of study entry
* Uncontrolled illness, physical disability, or other contraindication to aerobic exercise training including, but not limited to:

  * Acute myocardial Infarction (within 5 days of any planned study procedure)
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute (within 3 months) pulmonary embolus or pulmonary infarction
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Room air desaturation at rest =< 85%
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (ie infection, renal failure, thyrotoxicosis)
  * Mental impairment leading to inability to cooperate

NON-RANDOMIZED OBSERVATIONAL AND INTERVENTION COMPONENTS (ARM C):

The same exclusion criteria apply as above. Additionally,

• Should have no prior history of cancer, except for non-melanoma skin cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cardiopulmonary fitness (Arms A, C, and Observational groups only) | Up to 16 weeks
  Change in cardiopulmonary fitness as indicated by V02max (from CPET) will be compared across each arm. All analyses will employ the intention-to-treat (ITT) approach. Every attempt will be made to complete the week 16 follow-up assessment on all patients.

SECONDARY OUTCOMES:
Effect of aerobic training on general anxiety | At baseline and 16 weeks, 12 months and 24 months after start of intervention
  Subject will complete the State Trait Anxiety Inventory (STAI) for Adults survey to assess general anxiety scores. The survey measures state and trait anxiety, with 20 questions, and each question can be scored as 1-4 points. Higher scores indicate greater anxiety and the score range is 20-80.
Effect of aerobic training on specific prostate cancer anxiety | At baseline and 16 weeks, 12 months and 24 months after start of intervention
  Subjects will complete the Memorial Anxiety Scale for Prostate Cancer (MAXPC) survey to assess specific prostate cancer anxiety. Higher scores indicate greater anxiety and the fear of cancer recurrence score ranges from 0 to 12.
Adherence to active surveillance | At 12 months
  Adherence is measured by the proportion of patients in each study group that remain on active surveillance after 12 months follow-up.
Adherence to active surveillance | At 24 months
  Adherence is measured by the proportion of patients in each study group that remain on active surveillance after 24 months follow-up.
Messenger ribonucleic acid (mRNA) expression patterns and prognostic scores in tumor and surrounding stromal (normal) tissue | At baseline and 16 weeks after start of intervention
  Effect of aerobic training on mRNA expression patterns using the 1.4 million marker Affymetrix 1.0 Human Exon Array, in formalin-fixed paraffin-embedded (FFPE) prostate biopsy tissue taken before and after the intervention interval..

CONTACTS AND LOCATIONS:
Overall Officials: June Chan, Sc.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Blarigan EL, Kenfield SA, Olshen A, Panchal N, Encabo K, Tenggara I, Graff RE, Bang AS, Shinohara K, Cooperberg MR, Carroll PR, Jones LW, Winters-Stone K, Luke A, Chan JM. Effect of a Home-based Walking Intervention on Cardiopulmonary Fitness and Quality of Life Among Men with Prostate Cancer on Active Surveillance: The Active Surveillance Exercise Randomized Controlled Trial. Eur Urol Oncol. 2024 Jun;7(3):519-526. doi: 10.1016/j.euo.2023.10.012. Epub 2023 Oct 29. PMID 37907387
- See also: Link to Citation in European Urology Oncology (2024) — https://doi.org/10.1016/j.euo.2023.10.012

DOCUMENTS (1):
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT02435472/ICF_000.pdf